CLINICAL TRIAL: NCT00746057
Title: Evaluation of an Early Screening Test of Chronic Rejection and of Operational Tolerance by MicroArray in Renal Graft.
Brief Title: Evaluation of an Early Screening Test of Chronic Rejection and of Operational Tolerance by MicroArray in Renal Graft (Protocol DPRC Array)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of included patients is sufficient.
Sponsor: Nantes University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 06/2-E
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: First Cadaveric Renal Graft
Keywords: Renal graft; chronic rejection; tolerance; DNA chip; biopsy
MeSH Terms: interventions — Oligonucleotide Array Sequence Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Patients aged 18 to 65 years old receiving a first cadaveric renal graft.
  Interventions: Biological: DNA chip

INTERVENTIONS:
Biological: DNA chip — One biopsy is realized before graft, another biopsy is realized one year after graft and a blood sample is collected 3 months after graft to realize DNA chip. Blood samples are also collected at day 0, day 1, month 3, month 6 and month 12 to analyze biochemistry, proteinuria, haematology, creatinine clearance and immunology at day 0, month 3 and month 12.

SUMMARY:
The aim of the study is to explore the possibility to identify, at an early stage after a renal graft and from blood samples collected within first months after graft, a predictive transcriptional profile of long term occurence of graft operational tolerance or chronic rejection.

The aim of the study is to determine an early transcriptional profile of chronic rejection in the transcriptome of mononuclear blood cells. Validation and predictivity of transcriptional analysis will be based on graft function and graft histology one year after transplantation.The other aim is to determine an early transcriptional profile of operational tolerance in the same patients using a DNA chip dedicated including two lists of genes discriminating tolerant patients who are stopped immunosuppressant treatment for over a year.

To allow statistical analysis of 100 patients followed one year after graft, patients not assessable at one year due to early termination of study will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years old,
* Donor's age ≤ 60 years old,
* Patients receiving a first cadaveric renal graft,
* Patients taking immunosuppressant treatment including an induction with Simulect at day 0 and day 4, FK 506 (Prograf®) associated with Cellcept and steroids (for three months),
* Patients don't taking indispensable anticoagulant treatment.

Exclusion Criteria:

* Patient's age < 18 or > 65 years old,
* Donor's age ≥ 60 years old,
* Pregnant women or breast feeding women,
* Patients receiving a retransplantation, a kidney and pancreas graft or a graft from a living donor,
* Patients taking immunosuppressant treatment without FK 506 (Prograf®), Cellcept and steroids.
* Patients with coagulation troubles or taking indispensable anticoagulant treatment,
* No biopsy before graft.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2006-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Transcriptional profile (exhaustive DNAchip) on the blood at 3 months post transplantation. | 3 months

SECONDARY OUTCOMES:
Correlation of the transcriptional profile at 3 months after transplantation with histological features of the kidney graft at one year of follow-up. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul SOULILLOU, Professor, Principal Investigator — Nantes University Hospital; Magali GIRAL, Doctor, Study Chair — Nantes University Hospital; Maryvonne HOURMANT, Professor, Study Chair — Nantes University Hospital; Diego CANTAROVICH, Doctor, Study Chair — Nantes University Hospital; Jacques DANTAL, Professor, Study Chair — Nantes University Hospital; Gilles BLANCHO, Professor, Study Chair — Nantes University Hospital; Aurélie MEURETTE, Doctor, Study Chair — Nantes University Hospital; Marie LINO, Doctor, Study Chair — Nantes University Hospital; Georges MOURAD, Professor, Study Chair — University Hospital, Montpellier; Lionel ROSTAING, Professor, Study Chair — University Hospital, Toulouse; Dominique DURAND, Professor, Study Chair — University Hospital, Toulouse; Christophe LEGENDRE, Professor, Study Chair — AP-HP (Hôpital Necker); Michèle KESSLER, Professor, Study Chair — CHU NANCY; Emmanuel MORELON, Professor, Study Chair — Hospices Civils de Lyon; Sameh DAOUD, Doctor, Study Chair — Hospices Civils de Lyon; Cécile CHAUVET, Doctor, Study Chair — Hospices Civils de Lyon; Olivier THAUNAT, Doctor, Study Chair — Hospices Civils de Lyon; Jean-François SUBRA, Professor, Study Chair — University Hospital, Angers; François BAYLE, Doctor, Study Chair — University Hospital, Grenoble; Elisabeth CASSUTO, Doctor, Study Chair — CHU NICE
Locations (1):
- CHU de Nantes, Nantes, France